CLINICAL TRIAL: NCT06593067
Title: Skin Surface and Intradermal Temperature Responses to Heat Stress
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Crandall, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU_2024_0636
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hyperthermia
Keywords: Skin Temperature; Intradermal Temperature; Cooling Modalities
MeSH Terms: conditions — Hyperthermia | interventions — CCP110 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Intradermal Skin Temperature Needle in Intradermal Skin Layer (Active Comparator)
  Interventions: Other: Control; Other: Fan; Other: Fan and Water Spray; Other: Water Spray
- Intradermal Skin Temperature Needle on Skin Surface (Active Comparator)
  Interventions: Other: Control; Other: Fan; Other: Fan and Water Spray; Other: Water Spray
- Skin Temperature Thermistor on Skin Surface (Active Comparator)
  Interventions: Other: Control; Other: Fan; Other: Fan and Water Spray; Other: Water Spray

INTERVENTIONS:
Other: Control — Individuals will be exposed to a heated environment (41°C, 15% humidity) for a period of 15 minutes without a cooling modality.
Other: Fan — Individuals will be exposed to a heated environment (41°C, 15% humidity) for a period of 15 minutes with an electric fan as a cooling modality.
Other: Fan and Water Spray — Individuals will be exposed to a heated environment (41°C, 15% humidity) for a period of 15 minutes with an electric fan and water spray as cooling modalities.
Other: Water Spray — Individuals will be exposed to a heated environment (41°C, 15% humidity) for a period of 15 minutes with water spray as a cooling modality.

SUMMARY:
The purpose of this study is to compare surface and intradermal skin temperature responses to heat stress with and without evaporative and convective cooling.

DETAILED DESCRIPTION:
Humans have important thermoregulatory responses aimed at maintaining body temperature within a narrow range. These responses are driven in part by receptors located in the skin that monitor temperature changes and provide feedback to the central nervous system. Given that skin temperature can affect the physiological responses to heat stress, it is important to accurately measure skin temperature in response to heat stress with and without evaporative (i.e., sweat) and convective (i.e., air flow) cooling. Skin temperature is most often measured on the surface of the skin; however, this temperature can be influenced by other factors such as the local environment. It is unclear how the temperature of the skins surface compares to the temperature within the dermal layer of the skin.

The study team will directly compare skin surface and intradermal temperature responses to heat stress and determine whether these responses area altered by evaporative or convective cooling methods. To accomplish this objective, healthy adults will be exposed to ambient heat stress (no higher than 47°C) with and without evaporative (water sprayed on the skin) and convective (electric fan) cooling. Thermoregulatory responses, inclusive of skin surface and intradermal temperatures, will be assessed throughout the heat trial.

ELIGIBILITY:
Inclusion Criteria:

* Free of any significant underlying medical problems based upon a detailed medical history and physical exam.
* Normal resting electrocardiogram.

Exclusion Criteria:

* Known heart disease; other chronic medical conditions requiring regular medical therapy including cancer, diabetes, neurological diseases, and uncontrolled hypertension, etc.; as well as serious abnormalities detected on routine screening.
* Individuals who are pregnant, planning to become pregnant, or breastfeeding.
* Taking prescribed medications (such as beta blockers and non-dihydropyridine calcium channel blockers) or over-the-counter medications that have known influences on thermoregulatory response.
* Current smokers, as well as individuals who regularly smoked within the past 3 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Skin Temperature with Fan Only | 40 minutes into the heat intervention.
  Skin temperature will be measured from small temperature sensitive electrodes attached to the surface and intradermal layer of the skin of the participant with the fan cooling modality.
Skin Temperature with Fan and Water Spray | 60 minutes into the heat intervention.
  Skin temperature will be measured from small temperature sensitive electrodes attached to the surface and intradermal layer of the skin of the participant with both the fan and water spray cooling modalities.
Skin Temperature with Water Spray Only | 1 hour 20 minutes into the the heat intervention.
  Skin temperature will be measured from small temperature sensitive electrodes attached to the surface and intradermal layer of the skin of the participant with the water spray cooling modality.
Skin Temperature with No Cooling | 20 minutes into the heat intervention.
  Skin temperature will be measured from small temperature sensitive electrodes attached to the surface and intradermal layer of the skin of the participant during the heat intervention with no cooling.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Crandall, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No